CLINICAL TRIAL: NCT01591304
Title: Feasibility Study: Evaluation of the Safety and Effectiveness of the Ulthera® System for the Treatment of Moderate to Severe Facial Acne
Brief Title: Feasibility Study: Ulthera® System for the Treatment of Moderate to Severe Facial Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-116
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2014-12

CONDITIONS: Facial Acne
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Ulthera System Treatment provided using 1.5mm and 1.0mm transducers at 0.25J and 0.20J energy settings, respectively.
  Interventions: Device: Ulthera System Treatment
- Group B (Active Comparator): Ulthera System Treatment provided using 1.5mm and 1.0mm transducers, at 0.18J and 0.15J energy settings, respectively.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.

SUMMARY:
This study will evaluate the effectiveness of Ultherapy for the treatment of facial acne.

DETAILED DESCRIPTION:
Study subjects will be assigned to one of two treatment groups. Both treatment groups will receive treatment in the center of the forehead/temples, medial cheeks, and chin regions using the 1.5mm and 1.0mm transducers.

* For Group A, both the 1.5mm and 1.0mm transducers will be used at 0.25J energy setting and 0.20J energy setting, respectively.
* For Group B, both the 1.5mm and 1.0mm transducers will be used at 0.18J energy setting and 0.15J energy setting, respectively.

Subjects will receive 3 Ultherapy treatments administered 2 weeks apart. Subjects will be required to return for follow-up assessments at 14, 30, 60, 90 and 180 days following the third Ultherapy treatment. Pre- and post-treatment photos will be taken. In addition, pre- and post-treatment lesion counts and sebum measurements will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and older.
* Subject in good health.
* Presence of clinically-evident facial acne of moderate to severe severity with at least 20 inflammatory lesions and 20-100 noninflammatory lesions.

Exclusion Criteria:

* Presence of >2 nodular lesions in the areas to be treated.
* Presence of any cysts in the areas to be treated.
* Presence of an active systemic or local skin disease that may affect wound healing.
* Use of alcohol-based topical solutions or "exfoliating" agents within 1 week prior to study participation.
* History of frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
* History of keloid scar formation.
* Significant scarring in areas to be treated.
* Significant open facial wounds or lesions.
* Presence of a metal stent or implant in the facial area to be treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in facial acne | 60 days post-treatment
  Determined by a reduction in inflammatory and non-inflammatory lesion counts from baseline.

SECONDARY OUTCOMES:
Change from baseline in skin clarity | 180 days post-treatment
  Measured using a digital imaging system comparing baseline and post-treatment images.
Reduction of sebum production | 180 days post-treatment
  Assessments using a sebumeter will be performed comparing pre-treatment and post-treatment assessments.
Patient Satisfaction at 60 days | 60 day post-treatment
  Patient satisfaction as determined by completion of a patient satisfaction questionnaire.
Patient Satisfaction at 180 days | 180 Days post-treatment
  Patient satisfaction as determined by completion of patient satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Munavalli, M.D., Principal Investigator — Dermatology, Laser & Vein Specialists of the Carolinas
Locations (2):
- United States (2):
  - Multispecialty Aesthetic Clinical Research Organization, Woodland Hills, California
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina